CLINICAL TRIAL: NCT06261515
Title: Multi-omics Multi-specimens Evaluation of Oral-gut-systemic Profiles in Patients With Stage III-IV Periodontitis Pre- and After-therapy
Brief Title: Multi-omics Analysis of Oral-gut Microbial Profiles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perio-gut PRIN
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional periodontal treatment (Experimental): Periodontal treatment of stage III-IV periodontitis patients according to the guideline recommendation from the European Federation of Periodontology will be provided.
  Interventions: Procedure: Active periodontal treatment

INTERVENTIONS:
Procedure: Active periodontal treatment — Subgingival instrumentation with ultrasonic devices and curettes of all periodontal pockets; periodontal surgery if needed (residual probing pocket depths ≥ 6 mm).

SUMMARY:
Periodontitis is a chronic inflammatory disease of the tooth supporting structures induced by a dysbiosis in the oral and subgingival microenvironment of susceptible patients. The long-term swallowing of high doses of periodontal pathogenic microorganisms could induce a dysbiosis of the intestinal microbiota, favouring the establishment of an 'inflamed' microbiome in terms of composition and/or function. The present project is aimed at a better understanding of the etiopathogenetic correlation between periodontitis and intestinal dysbiosis, and aims to explore the hypothesis that periodontal treatment may influence the multi-omics profile on the oral-gut-systemic axis. 70 patients affected by stage III-IV periodontitis will be recruited, and treated by means of full-mouth scaling and root planing. Salivary, subgingival plaque, plasma and stool samples, together with a complete periodontal charting and a food diary will be collected and compared at baseline and after treatment. Age, gender and BMI-matched healthy individuals will be recruited as controls.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis Stage III or IV
* BMI between 20 and 29 kg/m2
* free diet
* presence of at least 20 teeth

Exclusion Criteria:

* systemic diseases (including diabetes, thyroid, liver, or kidney diseases)
* dietary allergies
* use of antibiotics or probiotics during the previous 90 days
* pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbial profile measured in stool samples | Baseline and 90 days
  Taxonomic variation of gut bacteria concentration after treatment assessed through shotgun metagenomics
Changes in oral microbial profile measured in saliva samples | Baseline and 90 days
  Taxonomic variation of salivary bacteria concentration after treatment assessed through shotgun metagenomics
Changes in oral microbial profile measured in subgingival plaque samples | Baseline and 90 days
  Taxonomic variation of subgingival bacteria concentration after treatment assessed through shotgun metagenomics

SECONDARY OUTCOMES:
Changes in oral-gut metabolome measured in stool samples | Baseline and 90 days
  Untargeted metabolic variation of oral-gut environment after treatment
Changes in oral-gut miRNAome measured in stool samples | Baseline and 90 days
  miRNA variation of oral-gut environment after treatment
Metabolic plasma changes | Baseline and 90 days
  Concentration of IL-1β, IL-6, IL-10, TNF-α, INF-γ, glucose, and cortisol released in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy